CLINICAL TRIAL: NCT04348929
Title: Birth Experience During COVID-19 Confinement (Confinement and Fostering Intrapartum Care)
Brief Title: Birth Experience During COVID-19 Confinement
Acronym: CONFINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, BERTHOLDT Charline, Principal Investigator (obstetrician-gynecologist), Central Hospital, Nancy, France
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2020-A00881-38
Record Dates: First submitted 2020-04-10; First posted 2020-04-16 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Postpartum Depression
Keywords: confinement; birth experience; covid-19
MeSH Terms: conditions — Depression, Postpartum; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Confinement group (Experimental): Delivery during covid-19 confinement period
  Interventions: Other: Self-administered questionnaires
- Control group (Other): Delivery after the withdrawal of all sanitary measures (mask, social distancing, limited visits during post-partum immediate)
  Interventions: Other: Self-administered questionnaires
- Epidemic group (Other): Delivery after confinement period and before the withdrawal of sanitary measures implemented (mask, social distancing, limited visits during post-partum immediate)
  Interventions: Other: Self-administered questionnaires

INTERVENTIONS:
Other: Self-administered questionnaires — Self-administered questionnaires once during the post-natal hospitalization and a second time 7 to 9 weeks after the delivery (at home)

SUMMARY:
Different studies have demonstrated that the absence of companionship during labor and childbirth may be responsible for a negative birth experience, an increased risk of postnatal depression and/or post traumatic stress disorders. These situation may also have a negative impact on mother-child interaction, on marital and family relationship and on the rate of maternal suicide in postpartum. However, these previous results cannot be extrapolated in the current context where the absence of the companionship is imposed by the confinement framework. The objective of the CONFINE study is to assess, for the first time, the birth experience of women in the context of limited social support in the immediate post-partum period due to confinement, as well as the associated over-risk of mental disorders, compared to a post-partum without social restriction.

DETAILED DESCRIPTION:
The primary objective is to compare, in immediate post-partum, the maternal sense of control during childbirth between a group of women who gave birth during confinement ("confinement" group) versus a group of women who gave birth after confinement but in the context of epidemic ("epidemic" group) versus a group of control women ("control" group; excluding confinement and context of epidemic).

The secondary objectives are:

1. To compare, at two months post-partum, the maternal sense of control during childbirth between the three groups.
2. To compare, at two months of post-partum, scoring of self-questionnaire Edinburg Postnatale Depression Scale (EPDS) for the post-natal depression between the three groups.
3. To compare at two months of post-partum, scoring of self-questionnaire Impact of Event Scale - Revised (IES-R) for posttraumatic stress disorder, between the three groups.
4. To compare, at two months of post-partum, the breastfeeding between the three groups.
5. To compare, at two months of post-partum, the quality of life (SF-12) between the three groups.
6. To compare the evolution of quality of life at two months of post-partum between the three groups.
7. To compare the rate of post-natal depression between the three groups.

ELIGIBILITY:
Inclusion Criteria:

* Woman who is >= 18 years old
* Woman having just given birth from 37 weeks of gestation (singleton pregnancy)
* Woman affiliated to a social security
* Woman with a level of understanding of written French sufficient to answer the questionnaires.
* Woman having received complete information on the organization of the research and having given her informed consent in written form.

Specific inclusion criteria according to the group For "confinement"group : Delivery during covid-19 confinement period

For "epidemic" group: Delivery after confinement period and before the withdrawal of sanitary measures implemented (mask, social distancing, limited visits during post-partum immediate)

For "control" group: Start of pregnancy after confinement and delivery after the withdrawal of all sanitary measures (mask, social distancing, limited visits during post-partum immediate)

Exclusion Criteria:

* Major mentioned in articles L.1121-6 and L-1121-8 of Health Public Code.
* Woman with psychiatric disorders such as depressive syndrome
* Woman considered positive for covid-19 and treated as such at the time of delivery (regardless of test result)
* Newborn with congenital abnormalities
* Stillbirth

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 927 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
"Labor Agentry Scale questionnaire" score in immediate post-partum (duration of hospital stay) | through study completion, an average of 16 months

SECONDARY OUTCOMES:
"Labor Agentry Scale questionnaire" score at two months after birth | through study completion, an average of 16 months
Edinburg Postnatale Depression Scale questionnaire" score at two months after birth | through study completion, an average of 16 months
  To detect suspicion of Post-Partum Depression
"Impact of Event Scale - Revised questionnaire" score at two months after birth | through study completion, an average of 16 months
  To detect suspicion of Post traumatic stress syndrome
Breastfeeding statement at two months after birth | through study completion, an average of 16 months
"SF-12 Quality of life questionnaire" score at two months after birth | through study completion, an average of 16 months
"SF-12 Quality of life questionnaire" score in immediate post-partum | through study completion, an average of 16 months
Diagnosis of post-natal depression (made by a specialist) | through study completion, an average of 16 months

CONTACTS AND LOCATIONS:
Overall Officials: Charline BERTHOLDT, Study Chair — Central Hospital, Nancy, France
Locations (1):
- Centre Hospitalier Régional Universitaire de Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: Yes
All data generated during this study will be made available via CIC-EC, CHRU Nancy, Nancy- FRANCE in accordance with protocol promotor. Data obtained from this study will be deposited at CIC-EC Nancy where they will be maintained for a minimum of 15 years.

REFERENCES:
- [Derived] Bertholdt C, Epstein J, Banasiak C, Ligier F, Dahlhoff S, Olieric MF, Mottet N, Beaumont M, Morel O. Birth experience during COVID-19 confinement (CONFINE): protocol for a multicentre prospective study. BMJ Open. 2020 Dec 10;10(12):e043057. doi: 10.1136/bmjopen-2020-043057. PMID 33303470